CLINICAL TRIAL: NCT03759600
Title: A Phase 2, Multicenter, Open-label, Single-arm Study to Evaluate the Safety and Efficacy of Niraparib in Japanese Patients With Advanced, Relapsed, High-grade Serous Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer Who Have Received 3 or 4 Previous Chemotherapy Regimens
Brief Title: Japan Phase 2 Study of Niraparib in Participants With Advanced, Relapsed Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Niraparib-2002; U1111-1222-4100 (Other: WHO); JapicCTI-184224 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
Keywords: Drug Therapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Niraparib 300 mg (Experimental): Niraparib 300 milligrams (mg), capsules, orally, once daily on Days 1 to 28 of each 28-day treatment cycle for up to 50 cycles.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib capsule

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of niraparib in participants with advanced, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer who have received 3 or 4 previous chemotherapy regimens.

DETAILED DESCRIPTION:
The drug being tested in this study is called niraparib. Niraparib is being tested to treat people who have the homologous recombination deficiency (HRD)-positive, advanced, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer. This study will look at the efficacy and safety of niraparib in Japanese participants.

The study will enroll approximately 16 participants. Participants will be enrolled to one group and after that will be asked to take niraparib capsules at the same time each day throughout the study:

- Niraparib 300 mg

This multi-center trial will be conducted in Japan. The overall time to participate in this study is approximately 23 months. Participants will make multiple visits to the clinic in the treatment period, and the post-treatment period including follow-up assessments after the last dose of the study drug.

ELIGIBILITY:
Inclusion Criteria

1. Japanese female participants aged 20 years or older on the day of signing informed consent.
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
3. Participants must agree to undergo tumor homologous recombination deficiency/deficient (HRD) testing, and this test result must show that participants have an HRD-positive tumor (defined by the presence of a deleterious or suspected deleterious breast cancer gene (BRCA) mutation or be positive for genomic instability) by the central laboratory selected by the sponsor.

   Note 1: The study HRD test result must be received prior to enrollment. The tumor sample may be submitted for HRD testing prior to the screening period (ie, within 40 days before Cycle 1 Day 1) if the consent has been obtained and it appears the participant is likely to meet other eligibility requirements.

   Note 2: If historic blood germline BRCA mutation (gBRCAmut) is detected by a prior gBRCAmut testing, then tumor HRD sample test results are not required prior to enrollment; however, HRD testing still needs to be performed.
4. Participants must have histologically diagnosed, relapsed, high-grade (Grade 2 or 3) serous epithelial ovarian, fallopian tube, or primary peritoneal cancer with recurrent disease and must have been previously treated with chemotherapy and have not experienced disease progression at least 6 months to the last chemotherapy containing platinum-based anticancer agents.
5. Participants must have completed 3 or 4 previous chemotherapy regimens. Participants must have completed their last chemotherapy regimen >4 weeks prior to treatment initiation.
6. Participants must have at least one measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) (v.1.1).
7. Participants must have performance status of ≤1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status Scale.
8. Participants must have adequate organ function as indicated by the following laboratory values:

   * Absolute neutrophil count (ANC) ≥1,500/μL.
   * Platelet count ≥150,000/μL.
   * Hemoglobin ≥10 g/dL.
   * Serum creatinine ≤1.5× institutional upper limit of normal (ULN) OR calculated creatinine clearance ≥50 mL/minute, using the Cockcroft-Gault equation.
   * Total bilirubin ≤1.5×ULN OR direct bilirubin ≤1×ULN.
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN unless liver metastases were present, in which case they had to be ≤5×ULN.
9. Participants must have formalin-fixed, paraffin-embedded tumor samples available from the primary or recurrent cancer or agree to undergo fresh biopsy prior to study treatment initiation.
10. Participants must be able to take oral medications.
11. Female participants of childbearing potential must be negative for pregnancy test (beta-human chorionic gonadotropin [β-hCG]) within 7 days prior to receiving the first dose of study treatment.
12. Female participants who:

    * Are postmenopausal for at least 1 year before the screening visit, OR
    * Are surgically sterile, OR
    * If they are of childbearing potential, agree to practice 1 highly effective method of contraception and 1 additional effective (barrier) method at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, OR
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods], condoms only, withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.)

Exclusion Criteria

1. Participants who have had palliative radiotherapy encompassing >20% of the bone marrow within 1 week of the first dose of study treatment.
2. Participants who have any known, persistent (>4 weeks), Grade ≥3 hematologic toxicity from last cancer therapy.
3. Participants who have any known, persistent (>4 weeks), Grade ≥3 fatigue during the last cancer therapy.
4. Participants who have received pelvic radiotherapy as treatment for primary or recurrent disease within 1 year of the first dose of study treatment.
5. Participants who have symptomatic, uncontrolled brain or leptomeningeal metastases.

   To be considered "controlled," central nervous system (CNS) disease must have undergone treatment (eg, radiation or chemotherapy) at least 1 month prior to study enrollment. The participant must not have had any new or progressive signs or symptoms related to the CNS disease and must have been taking a stable dose of steroids or no steroids (as long as these were started at least 4 weeks prior to enrollment] or no steroids). A scan to confirm the absence of brain metastases at baseline was not required. Participants with spinal cord compression might have been considered if they had received definitive treatment for this and evidence of clinically stable disease for 28 days.
6. Participants who have known hypersensitivity to the components of niraparib.
7. Participants who have had prior treatment with a known poly (adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitors.
8. Participant who have had treatment with any investigational products within 28 days or 5 half-lives (whichever was longer) before the first dose.
9. Participants who have had major surgery per Investigator judgment within 3 weeks of the first dose. Participant must have recovered from any effects of any major surgery.
10. Participants who have diagnosis, detection, or treatment of invasive second primary malignancy other than ovarian cancer ≤24 months prior to study enrollment (except basal or squamous cell carcinoma of the skin that was definitively treated). Note: Participants must not have any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML), irrespective of the time for disease history.
11. Participants who are considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days of the first dose) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, small bowel obstruction or other serious gastrointestinal disorder, or any psychiatric disorder that prohibits obtaining informed consent.
12. Participants who have received a transfusion (platelets or red blood cells) within 4 weeks of the first dose of study treatment.
13. Participants who have received a live virus or bacterial vaccines within 4 weeks of the first dose of study treatment.
14. Participants who have a history or current evidence of any condition, therapy, or lab abnormality (including active or uncontrolled myelosuppression [ie, anemia, leukopenia, neutropenia, thrombocytopenia]) that might confound the results of the study, interfere with the participant's participation throughout the study period, or study participation is not in the best interest of the participant.
15. Participants who are regular user (including "recreational use") of any illicit drugs at the time of signing informed consent or have a recent history (within the past year) of drug or alcohol abuse.
16. Participants who are pregnant or breast-feeding or expecting to conceive within the planned duration of the study.

    NOTE: If a breast-feeding woman discontinue breast-feeding, she may be enrolled in the study.
17. Participants who are immunocompromised (participants with splenectomy are allowed).
18. Participants who have known human immunodeficiency virus (HIV) positive.
19. Participants who have known hepatitis B surface antigen (HBsAg) positive, or known or suspected active hepatitis C virus (HCV) infection.

NOTE: Participants who are positive for hepatitis B core antibody (HBcAb) or hepatitis B surface antibody (HBsAb) can be enrolled but must have an undetectable hepatitis B virus (HBV) viral load. Participants who have positive hepatitis C virus antibody (HCVAb) must have an undetectable HCV viral load.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants with advanced, relapsed, high-grade serous epithelial ovarian, fallopian tube, or primary peritoneal cancer who have received 3 or 4 previous chemotherapy regimens.
Enrollment: 20 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (33):
- Japan (33):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Hirosaki University Hospital, Hirosaki, Aomori
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - The Jikei University Kashiwa Hospital, Kashiwa, Chiba
  - Shikoku Cancer Center, Matsuyama, Ehime
  - Ehime University Hospital, Tōon, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Kure Medical Center and Chugoku Cancer Center, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Kansai Rosai Hospital, Amagasaki, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Nippon Medical School Musashi Kosugi Hospital, Kawasaki, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Tohoku University Hospital, Sendai, Miyagi
  - University of the Ryukyus Hospital, Nakagami-gun, Okinawa
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital, Koto-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Chiba Cancer Center, Chiba
  - Chiba University Hospital, Chiba
  - Gifu University Hospital, Gifu
  - Kagoshima City Hospital, Kagoshima
  - Kyoto University Hospital, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Niigata University Medical & Dental Hospital, Niigata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Aoki D, Tabata T, Yanagida S, Nakamura T, Kondo E, Hamanishi J, Harano K, Hasegawa K, Hirasawa T, Hori K, Komiyama S, Matsuura M, Nakai H, Nakamura H, Sakata J, Takehara K, Takekuma M, Yokoyama Y, Kase Y, Sumino S, Soeda J, Kato A, Suri A, Okamoto A, Sugiyama T. Niraparib in Japanese patients with heavily pretreated, homologous recombination-deficient ovarian cancer: final results of a multicenter phase 2 study. J Gynecol Oncol. 2024 Sep;35(5):e114. doi: 10.3802/jgo.2024.35.e114. PMID 39251349
- [Derived] Okamoto A, Kondo E, Nakamura T, Yanagida S, Hamanishi J, Harano K, Hasegawa K, Hirasawa T, Hori K, Komiyama S, Matsuura M, Nakai H, Nakamura H, Sakata J, Tabata T, Takehara K, Takekuma M, Yokoyama Y, Kase Y, Sumino S, Soeda J, Suri A, Aoki D, Sugiyama T. Phase 2 single-arm study on the efficacy and safety of niraparib in Japanese patients with heavily pretreated, homologous recombination-deficient ovarian cancer. J Gynecol Oncol. 2021 Mar;32(2):e16. doi: 10.3802/jgo.2021.32.e16. Epub 2020 Dec 10. PMID 33327047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 17 investigative sites in Japan from 26 December 2018 to 28 December 2022.
Pre-assignment Details: Female participants with a diagnosis of advanced, relapsed, high-grade serious epithelial ovarian, fallopian tube, or primary peritoneal cancer who have received 3 or 4 prior lines of anti-cancer therapy and are platinum-sensitive to the last platinum-based therapy were enrolled to receive niraparib 300 mg in this study.
Period: Overall Study
Arm/Group | Niraparib 300 mg
Started | 20
Completed | 0
Not Completed | 20
Not completed — Adverse Event | 2
Not completed — Progressive Disease | 15
Not completed — Site Terminated by Sponsor | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least 1 dose of study drug and have measurable disease at Baseline.
Groups:
- Niraparib 300 mg: Niraparib 300 mg, capsules, orally, once daily on Days 1 to 28 of each 28-day treatment cycle for up to 50 cycles.
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 20
Time from First Diagnosis to First Dose [Median (Full Range); unit: years] — Duration in years from the date of first diagnosis to the date of start of study drug.
  years | 4.71 [2.5 to 16.2]
Primary Tumor Site [Count of Participants; unit: Participants] — Participant were categorized based on site of tumor are reported.
  Participants
    Ovarian | 13
    Primary Peritoneal | 5
    Fallopian Tube | 2
Cancer Stage (FIGO) at Time of Initial Diagnosis [Count of Participants; unit: Participants] — Cancer stage was based on federation of obstetrics and gynecology (FIGO) staging. Stages as I; Only in ovaries (IA: Only in endometrium, IC: Only in one or both ovaries or fallopian tubes); II: Has grown outside ovaries and is growing within pelvis (IIA: Limited to upper two-thirds of vagina, IIC: With positive peritoneal washings or ascites); III: Has spread outside pelvis into abdominal cavity or lymph nodes (IIIA: In lower third of vagina, has not grown into pelvic wall, IIIC: Larger than 2 cm on lining of abdomen and might also be in lymph nodes); IV: Has spread to other body organs.
  Participants
    IA | 1
    IC | 1
    IIB | 1
    IIC | 1
    IIIA | 1
    IIIC | 12
    IV | 3
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 155.9 (5.78)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 53.70 (9.701)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — Body Mass Index=weight (kg)/[height (m)^2]
  kilograms per meter square (kg/m^2) | 22.12 (4.074)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale was as follows: Grade 0: Fully active, able to perform all pre-disease activities without restriction; Grade 1: Restricted in physically strenuous activity, ambulatory, able to carry out light work; Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours; Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4: Completely disabled. Cannot carry on any self-care. Only categories with participants are reported.
  Participants
    0 | 15
    1 | 5
Number of Prior Lines of Chemotherapy [Count of Participants; unit: Participants] — Participants were categorized based on number of prior lines of chemotherapy as 3 and 4. Only categories with participants are reported.
  Participants
    3 | 12
    4 | 8
Prior Taxane [Count of Participants; unit: Participants]
  Participants Who Received Taxane | 20
Prior Bevacizumab [Count of Participants; unit: Participants]
  Participants Who Received Bevacizumab | 10
  Participants Who Did Not Receive Bevacizumab | 10
Prior Doxorubicin [Count of Participants; unit: Participants]
  Participants Who Received Doxorubicin | 9
  Participants Who Did Not Receive Doxorubicin | 11
Prior Liposomal Doxorubicin [Count of Participants; unit: Participants]
  Participants Who Did Not Receive Liposomal Doxorubicin | 20
Prior Gemcitabine [Count of Participants; unit: Participants]
  Participants Who Received Gemcitabine | 11
  Participants Who Did Not Receive Gemcitabine | 9
Duration between the End Date of the Last Chemotherapy Regimen and the First Dose of Study Treatment [Median (Full Range); unit: months] | 2.1 [1 to 27]
Duration between End Date of the Last Platinum-based Therapy and the First Dose of Study Treatment [Median (Full Range); unit: months] | 16.3 [1 to 36]
Prior Surgery/Procedure for Study Indication [Count of Participants; unit: Participants]
  Participants Who Had Prior Surgery | 20
Number of Prior Surgery/Procedure for Study Indication [Mean (Standard Deviation); unit: surgery] | 2.3 (1.34)
Prior Radiation Therapy Related to the Study Indication [Count of Participants; unit: Participants]
  Had Radiation Therapy | 2
  Had No Radiation Therapy | 18
Response to Last Platinum-based Therapy [Count of Participants; unit: Participants] — Response to last platinum-based therapy achieving complete response(CR), partial response(PR), progressive disease(PD) or Stable Disease(SD) per response evaluation criteria in solid tumors version 1.1(RECIST v.1.1) CR=disappearance of all target lesions and PR=atleast a 30% decrease in sum of diameters (SoD) of target lesions, taking as reference baseline SoD. PD=at least a 20% increase in SoD of target lesions, taking as reference smallest (nadir) SoD since (and including) baseline. SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  Participants
    Complete Response (CR) | 9
    Partial Response (PR) | 8
    Stable Disease (SD) | 2
    Unknown | 1
Time to Progression after the Last Platinum Therapy [Count of Participants; unit: Participants] — Participants with time to progression were categorized as 6-12 months and more than 12 months. Time to progression is defined as the time from the date of last administration of platinum therapy to the first documentation of disease progression.
  Participants
    6-12 Month | 12
    More Than 12 Month | 8
Ovarian Cancer Pathology Histological: Histologic Subtype [Count of Participants; unit: Participants] — Participants were categorized as serous, endometrioid, mucinous and other for histological subtype of ovarian cancer pathology.
  Participants
    Serous | 20
    Endometrioid | 0
    Mucinous | 0
    Other | 0
Ovarian Cancer Pathology Histological: Tumor Grade [Count of Participants; unit: Participants] — With regard to tumor grading, conventional FIGO/ gynecologic oncology group (GOG)/ world health organisation (WHO) criteria or two-tier system for grading ovarian serous carcinoma is used; participants with grade 3 tumors in FIGO/GOG/WHO criteria (among grade 1 as well differentiated, grade 2 as moderately differentiated, and grade 3 indicates poorly differentiated) or participants with high-grade tumors in two-tier system (among low-grade or high-grade) are reported.
  Participants
    Grade 2 | 1
    Grade 3 | 6
    High Grade | 13
Germline Breast Cancer (Gene) (BRCA1) Mutant [Count of Participants; unit: Participants] — Participants were categorized as positive, negative or unknown for mutation of BRCA1 gene. Only categories with participants are reported.
  Participants
    Without Mutant | 3
    Unknown | 17
Germline BRCA2 Mutant [Count of Participants; unit: Participants] — Participants were categorized as positive, negative or unknown for mutation of BRCA2 gene. Only categories with participants are reported.
  Participants
    Without Mutant | 3
    Unknown | 17
Homologous Recombination Deficiency/Deficient (HRD) Companion Diagnostic (CDx) Test Result [Count of Participants; unit: Participants] — Participants were categorized as positive, negative and unknown for HRD CDx test result. Only categories with participants are reported.
  Participants
    Positive | 20
Genomic Instability Status [Count of Participants; unit: Participants] — Participants were categorized as positive, negative and unknown for genomic instability status. Only categories with participants are reported.
  Participants
    Positive | 17
    Unknown | 3
Tumor BRCA1/BRCA2 Mutation Status [Count of Participants; unit: Participants] — Participants were categorized as positive, negative and unknown for BRCA1/BRCA2 mutation status.
  Participants
    Negative | 6
    Positive | 13
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants achieving CR or PR as assessed by the Investigator per RECIST v.1.1. CR was defined as disappearance of all target lesions and PR was defined as at least a 30% decrease in SoD of target lesions, taking as a reference the Baseline SoD.
Time Frame: Until disease progression or death (Up to 3.8 years)
Population: FAS included all participants who received at least 1 dose of study drug and have measurable disease at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
percentage of participants | 60.0

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documented CR or PR per RECIST v.1.1 to disease recurrence or objective disease progression whichever occurs first. CR was defined as disappearance of all target lesions and PR was defined as at least a 30% decrease in SoD of target lesions, taking as a reference the Baseline SoD.
Time Frame: Until disease progression or death (Up to 3.8 years)
Population: FAS included all participants who received at least 1 dose of study drug and have measurable disease at Baseline. Only Responders were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 12
months | 9.9 [3.9 to NA] — Upper limit of 95% confidence interval (CI) was not estimable due to low number of participants with events.

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants achieving CR, PR or SD as assessed by the Investigator per RECIST v.1.1. CR was defined as disappearance of all target lesions and PR was defined as at least a 30% decrease in SoD of target lesions, taking as a reference the Baseline SoD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the SoD of target lesions, taking as a reference the smallest (nadir) SoD since (and including) Baseline.
Time Frame: Until disease progression or death (Up to 3.8 years)
Population: FAS included all participants who received at least 1 dose of study drug and have measurable disease at Baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
percentage of participants | 90.0 [68.302 to 98.765]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug up to 30 days after the last dose or beginning of subsequent anticancer therapy, whichever came first (Up to 3.8 years)
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
Participants | 20

5. Secondary Outcome: Number of Participants With Grade 3 or Higher TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A TEAE was defined as an adverse event with an onset that occurs after receiving study drug. A severity grade was defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03. As per NCI-CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences; and Grade 5 scales as death related to AE.
Time Frame: as for outcome 4
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
Participants | 17

6. Secondary Outcome: Number of Participants With Serious TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) was any AE that results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event. TEAE was defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: as for outcome 4
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
Participants | 8

7. Secondary Outcome: Number of Participants With TEAEs Leading to Drug Discontinuation
Description: An AE was defined as any untoward medical occurrence in a participant who has enrolled in a study; it does not necessarily have a causal relationship with this treatment. A TEAE was defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: as for outcome 4
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
Participants | 2

8. Secondary Outcome: Number of Participants With TEAEs Leading to Dose Interruption
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
Participants | 15

9. Secondary Outcome: Number of Participants With TEAEs Leading to Dose Reduction
Description: as for outcome 7
Time Frame: as for outcome 4
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
Participants | 16

10. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time in months from the date of first study drug administration to the date of first documentation of PD or death as assessed by the RECIST v.1.1. Per RECIST 1.1, PD was defined as at least a 20% increase in the SoD of target lesions, taking as a reference the smallest (nadir) SoD since (and including) Baseline.
Time Frame: Until disease progression or death (Up to 3.8 years)
Population: FAS included all participants who received at least 1 dose of study drug and have measurable disease at Baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
months | 8.3 [5.6 to 13.8]

11. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time in months from the study enrollment to death due to any cause.
Time Frame: as for outcome 4
Population: FAS included all participants who received at least 1 dose of study drug and have measurable disease at Baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib 300 mg
Number analyzed (Participants) | 20
months | 24.9 [14.9 to NA] — Upper limit of 95% CI was not estimable due to low number of participants with events.

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose or beginning of subsequent anticancer therapy, whichever came first (Up to 3.8 years)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Groups:
- Niraparib 300mg: Niraparib 300 mg, capsules, orally, once daily on Days 1 to 28 of each 28-day treatment cycle for up to 50 cycles.
Arm/Group | Niraparib 300mg
All-Cause Mortality (participants affected / at risk) | 13/20
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib 300mg (N=20)
Anaemia (Blood and lymphatic system disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Platelet count decreased (Investigations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib 300mg (N=20)
Alanine aminotransferase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 14
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 4
Constipation (Gastrointestinal disorders) | 9
Decreased appetite (Metabolism and nutrition disorders) | 5
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Gamma-glutamyltransferase increased (Investigations) | 2
Headache (Nervous system disorders) | 7
Hypertension (Vascular disorders) | 6
Lymphocyte count decreased (Investigations) | 2
Malaise (General disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Nasopharyngitis (Infections and infestations) | 3
Nausea (Gastrointestinal disorders) | 12
Neuropathy peripheral (Nervous system disorders) | 2
Neutrophil count decreased (Investigations) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Palpitations (Cardiac disorders) | 4
Platelet count decreased (Investigations) | 10
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 8
Weight decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT03759600/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03759600/SAP_001.pdf